CLINICAL TRIAL: NCT03754764
Title: Phase I/II Study to Evaluate Treatment of Relapsed B-cell Acute Lymphoblastic Leukemia After CD19 CAR-T Adoptive Cellular Immunotherapy With CAR-T Cells Targeting CD38
Brief Title: A Feasibility and Safety Study of CD38 CAR-T Cell Immunotherapy for Relapsed B-cell Acute Lymphoblastic Leukemia After CD19 CAR-T Adoptive Cellular Immunotherapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Molecular & Immunological Department,Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-038
Record Dates: First submitted 2018-11-24; First posted 2018-11-27 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Relapsed B-cell Acute Lymphoblastic Leukemia After CD19 CAR-T ACI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Specificity CD38 CAR-T Cells — 1) Biological: Specificity CD38 CAR-T Cells 2) Day 0: 1-5x10e6/kg total dose .3) Other: Laboratory Biomarker Analysis

SUMMARY:
CD19-directed CAR-T cell therapy has shown promising results for the treatment of relapsed or refractory B-cell malignancies; however, a subset of patients relapse due to the loss of CD19 in tumor cells. CD38 CAR-T cells can recognize and kill the CD19 negative malignant cells through recognition of CD38. This is a phase 1/2 study designed to determine the safety of the gene-edited specificity CD38 CAR-T cells and the feasibility of making enough to treat patients with relapsed B-cell acute lymphoblastic leukemia after CD19 CAR-T adoptive cellular immunotherapy.

DETAILED DESCRIPTION:
1. PRIMARY OBJECTIVES:

   1. To evaluate the feasibility and safety of specificity CD38 CAR-T cells in patients with relapsed or refractory leukemia and lymphoma.
   2. To evaluate the duration of in vivo persistence of adoptively transferred T cells, and the phenotype of persisting T cells.

   Real Time polymerase chain receptor (RT-PCR) and Flow cytometry(FCM) analysis of PB,BM and lymph node will be used to detect and quantify survival of CD38 CAR-T cells over time.
2. SECONDARY OBJECTIVES:

   1. For patients with detectable disease, measure anti-tumor response due to specificity CD38 CAR-T cell infusions.
   2. The CAR-T cells will be administered by i.v. injection over 20-30 minutes as a using Day 0: 1-5x10e6/kg total dose on day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant
2. 12 Years to 70 Years (Child, Adult, Senior)
3. Patient with relapsed CD38+ B-cell acute lymphoblastic leukemia after CD19 CAR-T adoptive cellular immunotherapy
4. Estimated life expectancy ≥ 12 weeks (according to investigator's judgement)
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
6. Adequate organ function

Exclusion Criteria:

1. Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease
2. Diagnosis of Burkitt's leukemia/lymphoma according to WHO classification or chronic myelogenous leukemia lymphoid blast crisis
3. Richter's syndrome
4. Presence of Grade II-IV (Glucksberg) or B-D (IBMTR) acute or extensive chronic GVHD at the time of screening
5. Subjects with any autoimmune disease or any immune deficiency disease or other disease in need of immunosuppressive therapy
6. Severe active infection (uncomplicated urinary tract infections, bacterial pharyngitis is allowed), Prophylactic antibiotic, antiviral and antifungal treatment is permissible
7. Active hepatitis B, active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of screening
8. Patient has an investigational medicinal product within the last 30 days prior to screening
9. Previous treatment with investigational gene or cell therapy medicine products
10. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
11. Pregnant or nursing women

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-11-23 (Actual); Primary Completion 2022-11-23 (Estimated); Study Completion 2022-11-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe/Adverse Events as a Measure of Safety and Tolerability | 24 weeks
MTD of specificity CD38 CAR-T cells | 4 weeks
  The highest dose of specificity CD38 CAR-T cells that is estimated to result in defined Dose Limiting Toxicity (DLT) with the exception of allowable 'expected' AEs associated with the intravenous infusion of specificity CD38 CAR-T cells.
Copies numbers of CAR in peripheral blood(PB), bone marrow(BM)and lymph nodes | 24 weeks

SECONDARY OUTCOMES:
Six-month Objective response rate of complete remission and partial remission | 24 weeks
Six-month Overall survival | 24 weeks
Six-month Progression free survival | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Hematology Department of Chinese PLA, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided